CLINICAL TRIAL: NCT04056624
Title: Examining Validity and Sensitivity of Pressure-Mediated Reflection Spectroscopy as a Measure of Fruit and Vegetable Consumption in a Diverse Community
Brief Title: Examining Validity and Sensitivity of Pressure-Mediated Reflection Spectroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: University of Minnesota (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Stephanie Pitts, Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HL142544-01A1 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-08-14 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Dietary Habits; Diet, Healthy
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: First, investigators will examine the association (RS Device Validity) between RS-assessed skin carotenoids and the primary outcomes of objectively-measured plasma carotenoids and self-reported F&V consumption across four diverse groups: African-American/Black, Asian, White, and Hispanic/Latino. Then investigators will conduct a randomized controlled trial to define the relative skin carotenoid responses (RS Device Sensitivity) across racial-ethnic groups, in comparison with plasma carotenoid responses. Investigators will conduct a 6-week randomized controlled trial of a carotenoid-containing juice intervention [placebo control, low and high dose juice across 4 genetically-stratified racial-ethnic groups (n = 156).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): 1 x 6 ounces of carotenoid-containing juice (6 mg carotenoids/6 oz)
  Interventions: Dietary Supplement: High carotenoid juice
- High dose (Experimental): 2 x 6 ounces of carotenoid-containing juice (12 mg carotenoids/12 oz)
  Interventions: Dietary Supplement: High carotenoid juice
- Placebo (Placebo Comparator): 12 ounces of apple juice (negligible carotenoids 0.06 mg/12 oz)
  Interventions: Dietary Supplement: Placebo control - Apple juice

INTERVENTIONS:
Dietary Supplement: High carotenoid juice — Juice with high carotenoids
  Arms: High dose; Low dose
Dietary Supplement: Placebo control - Apple juice — Juice with negligible carotenoids
  Arms: Placebo

SUMMARY:
The central goal of this proposal is to examine validity and sensitivity of RS-assessed skin carotenoid status as a marker of F&V intake in a racially and ethnically diverse sample of individuals. First, investigators will examine the association (RS Device Validity) between RS-assessed skin carotenoids and the primary outcomes of objectively-measured plasma carotenoids and self-reported F&V consumption across four diverse groups: African-American/Black, Asian, White, and Hispanic/Latino (n=213). Then the investigators will conduct a randomized controlled trial to define the relative skin carotenoid responses (RS Device Sensitivity) across racial-ethnic groups, in comparison with plasma carotenoid responses. The investigators will conduct a 6-week randomized controlled trial of a carotenoid-containing juice intervention [placebo control, low and high dose juice (N=156). Finally, the genetic basis for racial/ethnic group differences in skin carotenoid responses to diet will be investigated through hypothesis-driven genomic analysis of participants from Aims 1 and 2.

DETAILED DESCRIPTION:
A diet rich in fruits and vegetables (F&Vs) is associated with lower risk of nutrition-related chronic diseases and all-cause mortality. Despite these benefits, the US population under-consumes F&Vs, with particularly low intake in disadvantaged populations. Low F&V intake results in higher rates of nutrition-related chronic disease among disadvantaged populations when compared with more advantaged populations. Detecting and addressing inadequate F&V intake in these populations is needed to reduce such disparities. Yet, there is still no commonly used predictive, objective measure of F&V intake for surveillance or determination of policy or intervention effectiveness. The current objective, "gold standard" marker of F&V intake is blood carotenoid concentration-an expensive, time-intensive, and invasive measurement. Traditional methods of self-reported dietary assessment are imprecise and have diminished utility in rural and disadvantaged populations due to low literacy, numeracy, and internet connectivity. In the past decade, skin carotenoid status assessed by non-invasive resonance Raman spectroscopy (RRS) has emerged as a promising biomarker of F&V intake. Reflection spectroscopy (RS) is an improvement over RRS, offering stronger signals, faster data acquisition, and greater portability in a commercially available device (Veggie Meter, Longevity Link Corporation). However, a hurdle impedes use of RS in scientific studies: to date, nearly all of the non-invasive skin carotenoid validation has been conducted in non-Hispanic whites, primarily by RRS. Therefore, it is critical to evaluate RS in racially and ethnically diverse populations. The central goal of this proposal is to examine validity and sensitivity of RS-assessed skin carotenoid status as a marker of F&V intake in a racially and ethnically diverse sample of individuals. First, the investigators will examine the association (RS Device Validity) between RS-assessed skin carotenoids and the primary outcomes of objectively-measured plasma carotenoids and self-reported F&V consumption across four diverse groups: African-American/Black, Asian, White, and Hispanic/Latino (target n = 320 but due to Covid-19, N=213). Then the investigators will conduct a randomized controlled trial to define the relative skin carotenoid responses (RS Device Sensitivity) across racial-ethnic groups, in comparison with plasma carotenoid responses. The investigators will conduct an 6-week randomized controlled trial of a carotenoid-containing juice intervention [placebo control, low and high dose juice across 4 genetically-stratified racial-ethnic groups (goal n = 156). Finally, the genetic basis for racial/ethnic group differences in skin carotenoid responses to diet will be investigated through hypothesis-driven genomic analysis of participants from Aims 1 and 2. The results of this study will prepare RS for mass deployment in population surveillance studies and community-based intervention trials, ultimately leading to more accurate determination of the most effective strategies to reduce health disparities related to low F&V intake in the United States and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as one of the racial/ethnic groups of focus
* Read/speak English
* Between 18 and 65 years of age
* BMI 18.5-34.9 kg/m2
* Non-pregnant
* Non-lactating
* Healthy (no chronic disease)
* Not taking lipid-altering medication (medicines that lower cholesterol or triglycerides)
* Weight stable (have not gained or lost more than 15 pounds in the last 3 months).

Exclusion Criteria:

* Not of one of the four racial/ethnic groups of focus
* Not able to read/speak English
* Under 18 years of age or over 65 years of age, do not
* BMI less than 18.5 or more than 34.9 kg/m2
* Pregnant (or have been pregnant in the last 6 weeks)
* Lactating
* High blood sugar ( ≥126 mg/dl)
* Chronic disease such as cardiovascular disease, diabetes, chronic kidney disease, diabetes cancer other than non-melanoma skin cancer (within the last 5 years), or other weight-related chronic diseases.
* Taking medication that lowers cholesterol or triglycerides Diagnosed with/ treated for Crohn's disease.
* Not weight stable (gained or lost more than 15 pounds in the last three months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Jilcott Pitts, PhD, Principal Investigator — East Carolina University
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - East Carolina University, Greenville, North Carolina
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available to share with other investigators 12 months after study completion.
Access Criteria: Researchers must submit a plan for analysis, obtain Institutional Review Board approval and be approved by study investigators before data are released.

REFERENCES:
- [Derived] Jilcott Pitts SB, Wu Q, Laska MN, Moran NE. Two Spectroscopy Devices Can Approximate Fruit and Vegetable Intake in a Racially and Ethnically Diverse Sample. Curr Dev Nutr. 2025 Jun 4;9(7):107482. doi: 10.1016/j.cdnut.2025.107482. eCollection 2025 Jul. PMID 40654376
- [Derived] Jilcott Pitts SB, Wu Q, Moran NE, Laska MN, Harnack L. Examining Potential Modifiers of Human Skin and Plasma Carotenoid Responses in a Randomized Trial of a Carotenoid-Containing Juice Intervention. J Nutr. 2023 Nov;153(11):3287-3294. doi: 10.1016/j.tjnut.2023.09.014. Epub 2023 Sep 23. PMID 37742797
- [Derived] Jilcott Pitts S, Moran NE, Laska MN, Wu Q, Harnack L, Moe S, Carr-Manthe P, Gates E, Chang J, Zaidi Y, Gelineau A, Berg L, Craft NE. Reflection Spectroscopy-Assessed Skin Carotenoids Are Sensitive to Change in Carotenoid Intake in a 6-Week Randomized Controlled Feeding Trial in a Racially/Ethnically Diverse Sample. J Nutr. 2023 Apr;153(4):1133-1142. doi: 10.1016/j.tjnut.2023.02.017. Epub 2023 Feb 18. PMID 36804322

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose: 1 x 6 ounces of carotenoid-containing juice (4 mg carotenoids/6 oz)
  High carotenoid juice: Juice with high carotenoids
- High Dose: 2 x 6 ounces of carotenoid-containing juice (8 mg carotenoids/12 oz)
  High carotenoid juice: Juice with high carotenoids
- Placebo: 6 ounces of apple juice (negligible carotenoids 0.03 mg/6oz)
  Placebo control - Apple juice: Juice with negligible carotenoids
Period: Overall Study
Arm/Group | Low Dose | High Dose | Placebo
Started | 53 | 56 | 53
Completed | 52 | 54 | 52
Not Completed | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 6 ounces of apple juice (negligible carotenoids 0.03 mg/6 oz)
  Placebo control - Apple juice: Juice with negligible carotenoids
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 53 | 56 | 53 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (11.8) | 32.5 (11.4) | 31.3 (10.1) | 32.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 36 | 83
  Male | 33 | 29 | 17 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 14 | 13 | 13 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 15 | 13 | 41
  White | 14 | 15 | 15 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 13 | 12 | 37
Skin Carotenoid Level [Mean (Standard Deviation); unit: units on a scale] — Skin carotenoid level is a number from 0 to 800 that approximates carotenoids in the skin. The Veggie Meter device uses pressure mediated reflection spectroscopy to assess skin carotenoid level in the fingertip. Skin carotenoid levels are positively correlated with fruit and vegetable intake. A higher score generally indicates more fruit and vegetable intake, which is thought to be a better outcome.
  units on a scale | 310.8 (101.7) | 290.2 (89.1) | 293.6 (100.9) | 298.0 (97.1)

OUTCOME MEASURES:

1. Primary Outcome: 3-week Change in Skin Carotenoid Status
Description: Skin carotenoid level is a number from 0 to 800 that approximates carotenoids in the skin. The Veggie Meter device uses pressure mediated reflection spectroscopy to assess skin carotenoid level in the fingertip. Skin carotenoid levels are positively correlated with fruit and vegetable intake. A higher score generally indicates more fruit and vegetable intake, which is thought to be a better outcome. The primary outcome was change in skin carotenoid levels calculated by the skin carotenoid value at 3 weeks minus the value at baseline.
Time Frame: Change in skin carotenoid status from baseline to 3 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 52 | 54 | 52
units on a scale | 28.0 [15.6 to 40.5] | 62.3 [49.6 to 74.9] | 9.34 [-1.14 to 19.8]

2. Primary Outcome: 6-week Change in Skin Carotenoid Status
Description: Skin carotenoid level is a number from 0 to 800 that approximates carotenoids in the skin. The Veggie Meter device uses pressure mediated reflection spectroscopy to assess skin carotenoid level in the fingertip. Skin carotenoid levels are positively correlated with fruit and vegetable intake. A higher score generally indicates more fruit and vegetable intake, which is thought to be a better outcome. The primary outcome was change in skin carotenoid levels calculated by the value at 6 weeks minus the value at baseline.
Time Frame: Change in skin carotenoid status from baseline to 6 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 52 | 54 | 52
units on a scale | 59.0 [42.0 to 76.1] | 123 [105 to 141] | 11.9 [0.16 to 23.6]

ADVERSE EVENTS:
Time Frame: The time frame was through 6-weeks, or over the study duration for each participant.
Arm/Group | Low Dose | High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/54 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/54 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/54 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT04056624/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT04056624/ICF_000.pdf